CLINICAL TRIAL: NCT02460107
Title: Botulinum Toxin Type A for Neuropathic Pain in Patients With Diabetic Peripheral Polyneuropathy
Acronym: BTXADMPPNP
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrolling failure (lack of participants)
Sponsor: Catholic University of Korea Saint Paul's Hospital (Other)
Collaborators: Medy-Tox (Industry)
Responsible Party: Principal Investigator, Myung Eun Chung, MD, PhD, Catholic University of Korea Saint Paul's Hospital, Catholic University of Korea Saint Paul's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CatholicUKSPH
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal saline (Placebo Comparator): Normal saline
  Interventions: Other: Normal saline
- Botulinum toxin type A 50U (Active Comparator): Botulinum toxin 50U
  Interventions: Biological: Botulinum toxin type A
- Botulinum toxin type A 100U (Active Comparator): Botulinum toxin 100U
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A
  Arms: Botulinum toxin type A 100U; Botulinum toxin type A 50U
Other: Normal saline — Placebo
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine whether botulinum toxin A is effective in the treatment of neuropathic pain in patients with diabetic peripheral polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* • more than twenty years of age

  * patients should have 4 or more items positive among the 10 items of the DN4 questionnaire.
  * persistence of neuropathic pain for more than three months or remission and recurrence of neuropathic pain for more than six months
  * a pain score of 4 or more on the numeric rating scale

Exclusion Criteria:

* • neuropathic pain caused by confounding factors other than diabetic neuropathic pain

  * contraindicated for botulinum toxin type A
  * a change in pain medication one month prior to study enrollment
  * a condition involving neuromuscular junction (Ex. Eaton Lambert disease, myasthenia gravis)
  * person who received botulinum toxin type A within three months prior to study enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity using numeric rating scale | 4 weeks after intervention

SECONDARY OUTCOMES:
Pain intensity using numeric rating scale | 1, 8, 12, 24 weeks after intervention
Quality of life using WHOQOL | 4,8,12 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, The Catholic University of Korea, Seoul, South Korea